CLINICAL TRIAL: NCT05392582
Title: MicroRNA Regulation of Chronic Inflammation During Aging
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Micah Drummond, Professor, University of Utah
Other Study IDs: 153158
Record Dates: First submitted 2022-05-20; First posted 2022-05-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Chronic Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young: Young healthy adult participants
- Older: Older healthy adult participants

SUMMARY:
This is an observational study enrolling healthy individuals aged 18-35 and 65y and older to determine the health of immune cells in the blood and how these cells create inflammation and effect health as we age. It is hoped that once the nature of this relationship has been discovered we can more effectively design therapies to reduce this inflammation.

The enrollment goal is 40 participants. The study will occur over the course of 1 month which will include a screening visit and a second visit where the participants will undergo an oral glucose tolerance test, blood draws and leg strength & exercise tests.

DETAILED DESCRIPTION:
We will recruit healthy, non-obese (<30kg/m2 BMI) younger (N=20; 18-35y) and older (N=20; >65y) male and female participants (as determined by sample size calculation) in the Salt Lake City area.

1. VISIT 1 (Screening, visit duration: 1 hour): Once the participant is identified, they will be scheduled for a screening visit at the CTSI (421 Wakara Way) to see if they meet incl/excl criteria and to sign an informed consent document. As part of the visit, Upon arrival, we will gather basic health information such as height, weight, blood pressure, and heart rate.

   * Participant will undergo the following procedures: a blood screening (30ml of blood collected)
   * For older cohort: The clinical frailty scale (CFS) and Mini-Cog© cognitive assessment
2. VISIT 2 (visit duration: 3 hours) Following a 10h fast, participants will arrive in the morning. Upon arrival, we may gather basic health information from the participant such as height, weight, blood pressure, and heart rate. The procedures to take place at this visit are as follows:

   * 120 mL serum blood sample collection. Samples will be used to identify the immune cell populations in the blood, regulators of these immune cells and how these cells function.
   * Oral glucose tolerance test (OGTT)- participants will be asked to complete a test to determine their blood sugar levels. We will ask them to drink a sugary liquid (glucola) and then rest quietly while we measure changes in their blood sugar levels. We will draw 20 ml of blood during this test (~1 tablespoon). OGTT will take approximately 2hours.
   * Leg strength tests at the SMERF facility. Isometric strength will be assessed in both legs with a maximal voluntary isometric contraction effort developed by the knee extensors (quadriceps) on a isokinetic dynamometer. For lower extremity extension power testing a Nottingham power rig will be used. Total time for these tests will take 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 - 35y; 65y and older
2. BMI: <30 kg/m2
3. Ability to sign informed consent
4. For older participant group: Clinical Frailty Scale score < 3 and Mini-Cog score > 3
5. Good general medical health, ambulatory and in independent living setting

Exclusion Criteria:

* History of cardiovascular disease (e.g., CHF, CAD, MI, CVA)
* History of endocrine or metabolic disease such as hypo/hyperthyroidism and diabetes (Treated hypo/hyperthyroid for at least 6 months will be permitted)
* History of kidney disease or failure (CKD > stage 4)
* History of vascular disease
* Uncontrolled hypertension - Elevated systolic pressure >150 or a diastolic blood pressure > 100
* Cancer or history of successfully treated cancer (less than 1 year) other than basal cell carcinoma
* Chronic systemic corticosteroid use (≥ 2 weeks) within 4 weeks of enrollment and for study duration (intra-articular/topical/inhaled therapeutic or physiologic doses of corticosteroids will be permitted)
* Chronic anti-inflammatory medication use (≥ 2 weeks) within 4 weeks of enrollment
* Chronic inflammatory conditions (e.g., Rheumatoid Arthritis, Crohn's, fibromyalgia, lupus, colitis) HIV, Hepatitis B and C
* History of stroke with motor disability
* A recent history (<12 months) of GI bleed
* History of liver disease or AST/ALT 2 times above the normal limit
* History of respiratory disease (acute upper respiratory infection, history of chronic lung disease)
* Current smokers or current tobacco use
* Current pregnancy as determined by positive pregnancy test
* Any staff members who report directly to the principal investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy young and older adults
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Inflammation | Determined in older adults and in younger adults at a single visit (baseline).
  IL-6 levels

CONTACTS AND LOCATIONS:
Overall Officials: Micah Drummond, Principal Investigator — The University of Utah
Locations (1):
- The University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
No plan has been put into place